CLINICAL TRIAL: NCT06696950
Title: Effects of Multimodal Gait Training With and Without Rhythmic Auditory Stimulation on Coordination, Gait and Risk of Fall in Chronic Stroke Patients
Brief Title: Multimodal Gait Training With and Without Rhythmic Auditory Stimulation in Chronic Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0202
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Chronic Stroke Patients
Keywords: Chronic Stroke; Gate Training; Multimodal; Rhythmic auditory stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A received Multimodal gait training with Rhythmic auditory stimulation
  Interventions: Other: Mutimodal gait training includes unilateral step training, inclined treadmill training, over ground training with rhythmic auditory stimulation
- Group B (Experimental): Group B Multimodal Gait training without rhythmic auditory stimulation
  Interventions: Other: Multimodal gait training

INTERVENTIONS:
Other: Mutimodal gait training includes unilateral step training, inclined treadmill training, over ground training with rhythmic auditory stimulation — Unilateral step training, inclined treadmill training, over ground training, repetitive isochronous pulses via metronome
  Arms: Group A
Other: Multimodal gait training — Unilateral step training, inclined treadmill training, over ground training,
  Arms: Group B

SUMMARY:
The primary goal of this randomized clinical trial is to investigate the efficacy of multimodal gait training, with and without rhythmic auditory stimulation, in improving gait, coordination and reducing fall risk in individuals with chronic stroke This clinical trial features two distinct groups 42 participants were randomly divided into two groups of 21. Group A will receive Multimodal gait training along with rhythmic auditory stimulation while Group B will receive only multimodal gait training

Participants will:

* Take 12 sessions of the MMGT program over six weeks
* With each session lasting 45 minutes, including 10-minute rest breaks.

ELIGIBILITY:
Inclusion Criteria:

* Participants of age between 45 and 70 year
* Participants of both genders were included.
* Participants who were able to walk independently indoors without walking aid
* Participants were included if they had lower limb motor impairment (Fugl-Meyer Assessment lower extremity (FMLE) score less than score less than 34
* Participants with stroke lasting longer than six months
* Participants with Mini-Mental Status Examination score 24 or more than 24
* Participants with the capability to keep in sitting position for 30 minutes
* Participants with the history of fall in the past year
* Participants with no visual or auditory impairments that would interfere with the training

Exclusion Criteria:

* Participants with respiratory problems.
* Participants with any orthopedic condition.
* Participants with aphasia that impeded communication.
* Participants with have severe cardiac disease.
* Participants with resistant hypertension despite use of medication (average systolic blood pressure ≥ 140 mmHg or average diastolic blood pressure ≥ 90 mmHg measured over 7 days)
* Participants with presence of non-healing ulcers in the lower limbs, and osteoporosis

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
LOWER EXTREMITY MOTOR COORDINATON TEST (LEMCOT) | 6 weeks
  The Lower Extremity Motor Coordination test (LEMCOT) is a clinically useful performance-based test to assess coordination improvements of lower limb in post-stroke individuals
Dynamic gait index (DGI) | 6 weeks
  The dynamic gait index is a comprehensive clinical assessment performance based tool used designed to evaluate gait-related task such as dynamic balance, gait and risk of fall in older adults with various neurological conditions
Fall Efficacy Scale-International (FES-I) | 6 weeks
  Fall efficacy scale-international (FES- I) is a standardized, short and easy to administer tool evaluates fear of falling and measures concerns about falling

CONTACTS AND LOCATIONS:
Overall Officials: Binish Afzal, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- Allama Iqbal Memorial Hospital, Islam teaching hospital, National Bone joint Hospital, Amra Medical Center, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No